CLINICAL TRIAL: NCT05106270
Title: The Impact of Atrial Pressure Change Before and After One-stop Procedure Combining Catheter Ablation and Left Atrial Appendage Closure on the Prognosis of Patients With Atrial Fibrillation
Brief Title: The Impact of Atrial Pressure Change Before and After Combined Procedure
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief physician, Shanghai 10th People's Hospital
Other Study IDs: APPREANCE-AF
Record Dates: First submitted 2021-09-20; First posted 2021-11-03 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Left atrial pressure; combined procedure; Catheter ablation; Left atrial appendage closure; Cardiac function
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Besides routine peripheral blood sample for clinical use, intra-atrial blood sample 1-2ml are collected for biochemical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined procedure: The whole cohort underwent combining procedure of catheter ablation and left atrial appendage closure, atrial pressure was measured before and after pulmonary vein isolation, and after left atrial appendage closure.
  Interventions: Diagnostic Test: Atrial pressure measurement using transseptal puncture sheath

INTERVENTIONS:
Diagnostic Test: Atrial pressure measurement using transseptal puncture sheath — both left and right atrial pressure was measured using transseptal puncture sheath before and after combined procedure

SUMMARY:
One-stop procedure combining catheter ablation (CA) and left atrial appendage closure (LAAC) has been a feasible treatment for patients with atrial fibrillation at high risk of stroke and/or bleeding. Although it could achieve considerable rhythm control and stroke prophylaxis, a number of patients has experienced progressive heart failure after the procedure. Notably, previous studies indicate that both pulmonary vein isolation by CA and LAAC could significantly increase left atrial pressure, while currently no study has investigated left atrial pressure change in patients underwent combined procedure. The investigators hypothesise that combined procedure would significantly increase left atrial pressure and subsequently deteriorate cardiac function. Therefore, the investigators aim to measure the left and right atrial pressure change before and after CA and LAAC in combined procedure, and investigate the influence of the pressure change on clinical outcomes.

DETAILED DESCRIPTION:
1. Study aim. This study was designed to measure the left and right atrial pressure change before and after catheter ablation (CA) and left atrial appendage closure (LAAC) combining procedure, and investigate the influence of the pressure change on clinical outcomes.
2. Subject selection. This study is designed to recruit patients diagnosed with atrial fibrillation and planned to undergo combined procedure. Primary inclusion criteria are:

   i. Atrial fibrillation recorded by 12-lead ECG or Holter that last for longer than 30 seconds within the preceding 6 months; ii. Eligible for left atrial appendage closure, that meet at least one of the followings:
   1. At high risk of stroke (CHA2DS2-VASc score≥3 in female, ≥2 in male) and/or bleeding (HAS-BLED score≥3);
   2. Contraindicated to oral anticoagulation (OAC);
   3. Refused OAC treatment albeit comprehensively informed of the necessity and benefits of OAC treatment.
3. Procedure detail. All the patients recruited is planned to undergo combined procedure. CA is performed before LAAC. For CA, the energy source is optional (either radiofrequency or cryoenergy). And ablation should be performed for pulmonary vein isolation only. For LAAC, the occluder type is optional (either plug or pacifier occluder), and intracardiac echocardiography or transesophageal echocardiography (TEE) is optional.

   For atrial pressure measurement, right atrial pressure should be measured before transseptal puncture and after combined procedure is accomplished. Left atrial pressure should be measured at 3 timepoints: after transseptal puncture, after pulmonary vein isolation and after LAAC. Atrial pressure is measured via Swartz transseptal puncture sheath. And at each timepoint, atrial pressure should be recorded at 1min, 3min, and 5min after the placement of the sheath.
4. Follow-up. study endpoint includes a primary composite endpoint of rehospitalization due to heart failure and death due to cardiovascular disease, and secondary endpoints including: 1. all-cause mortality 2. major cardiovascular adverse event 3. rehospitalization due to cardiovascular diseases 4. recurrence of atrial arrhythmia 5. stoke/transient ischemic attack 6. echocardiographic measurement 7. quality of life evaluation 8. cardiac function evaluation 9. evaluation of left atrial appendage closure. Patients are required to have outpatient follow-up at 3rd month, 12th month, and every year since then. The anti-thromboembolic regimen should follow: 3-month OAC treatment and 3-month double anti-platelet therapy and lifelong single anti-platelet therapy. For LAAC follow-up, either TEE or CTA is scheduled to perform in the 3rd month after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation recorded by 12-lead ECG or Holter that last for longer than 30 seconds within the preceding 6 months;
* Eligible for left atrial appendage closure, that meet at least one of the followings:

  1. At high risk of stroke (CHA2DS2-VASc score≥3 in female, ≥2 in male) and/or bleeding (HAS-BLED score≥3);
  2. Contraindicated to oral anticoagulation (OAC);
  3. Refused OAC treatment albeit comprehensively informed of the necessity and benefits of OAC treatment.
* Capable of understanding and signing the informed consent form.
* Aged over 18 years.

Exclusion Criteria:

* Reversible causes of atrial fibrillation, including thyroid disorders, recent major surgery, trauma, acute alcoholic intoxication;
* Concomitant arrhythmia including atrial flutter, ventricular tachycardia;
* A previous history of atrial fibrillation surgery (MAZE surgery) or catheter ablation;
* A previous history of cardiac surgery including any valvular replacement, septal repair;
* A recent history of major cardiovascular disease within 3 months, including acute myocardial infarction, ventricular fibrillation;
* A history of congenital heart disease;
* A previous history of atrioventricular node ablation;
* A history of lobectomy due to any medical condition;
* Complicated by other diseases with life expectation <1 year;
* Women with childbearing potential;
* Participated in other interventional clinical trials that might affect prognosis;
* Unable to understand or give informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed to investigate the change of atrial pressure before and after combined procedure of catheter ablation and left atrial appendage closure, and evaluate its influence on prognosis. This study aims to recruit patients diagnosed with atrial fibrillation who are eligible for combined procedure. Patients with paroxysmal, persistent, or longstanding persistent AF are included, whether it is new-onset or drug refractory.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint | From date of inclusion until the date of first documented rehospitalization due to heart failure or date of death due to cardiovascular disease, whichever came first, assessed up to 60 months
  Rehospitalization due to heart failure and death due to cardiovascular disease

SECONDARY OUTCOMES:
All-cause mortality | From date of inclusion until the date of documented death of any reason, assessed up to 60 months
  death of any reason
Major cardiovascular adverse event | From date of inclusion until the date of first documented cardiovascular events mentioned above, assessed up to 60 months
  cardiovascular events including myocardial infarction, malignant arrhythmia, acute heart failure, cardiac tamponade.
Rehospitalization due to cardiovascular diseases | From date of inclusion until the date of first documented rehospitalization due to cardiovascular diseases, assessed up to 60 months
  Rehospitalization due to any cardiovascular diseases
Early recurrence of atrial arrhythmia | From time of completion of combined procedure until the third month since the procedure
  Atrial tachycardia, atrial flutter, or atrial fibrillation that last for longer than 15 seconds recorded by ECG or Holter
Recurrence of atrial arrhythmia | From the third month since the procedure until the date of recurrence of atrial arrhythmia as described above, assessed up to 60 months
  Atrial tachycardia, atrial flutter, or atrial fibrillation that last for longer than 15 seconds recorded by ECG or Holter
Stoke/transient ischemic attack | From date of inclusion until the date of first documented stoke/transient ischemic attack, assessed up to 60 months
  Cerebral infarction, intracranial hemorrhage, or transient ischemic attack confirmed by CT/MRI
Change from baseline echocardiographic measurement at 3 months | 3 months after combined procedure
  Echocardiographic measured left atrial parameters including left atrial volume, left atrial volume index, e, e' and left ventricle parameters including left ventricular ejection fraction, left ventricle systolic and diastolic diameter.
Change from baseline echocardiographic measurement at 1 year | 1 year after combined procedure
  Echocardiographic measured left atrial parameters including left atrial volume, left atrial volume index, e, e' and left ventricle parameters including left ventricular ejection fraction, left ventricle systolic and diastolic diameter.
Change from baseline echocardiographic measurement at 5 years | 5 years after combined procedure
  Echocardiographic measured left atrial parameters including left atrial volume, left atrial volume index, e, e' and left ventricle parameters including left ventricular ejection fraction, left ventricle systolic and diastolic diameter.
Change from baseline quality of life evaluation at 3 months | 3 months after combined procedure
  EQ-5D questionnaire evaluation of quality of life
Change from baseline quality of life evaluation at 1 year | 1 year after combined procedure
  EQ-5D questionnaire evaluation of quality of life
Change from baseline quality of life evaluation at 5 years | 5 years after combined procedure
  EQ-5D questionnaire evaluation of quality of life
Change from baseline walking distance of 6-min walk test at 3 months | 3 months after combined procedure
  Maximum walking distance measured from 6-min walk test
Change from baseline walking distance of 6-min walk test at 1 year | 1 year after combined procedure
  Maximum walking distance measured from 6-min walk test
Change from baseline walking distance of 6-min walk test at 5 years | 5 years after combined procedure
  Maximum walking distance measured from 6-min walk test
Evaluation of left atrial appendage closure at 3 months | 3 months after combined procedure
  Either transesophageal echocardiography or CTA evaluation of occluder position, residual flow, presence of thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided